CLINICAL TRIAL: NCT05429502
Title: Phase I/II Multicenter Study to Assess Efficacy and Safety of Ribociclib (LEE011) in Combination With Topotecan and Temozolomide (TOTEM) in Pediatric Patients With Relapsed or Refractory Neuroblastoma and Other Solid Tumors
Brief Title: Study of Efficacy and Safety of Ribociclib (LEE011) in Combination With Topotecan and Temozolomide (TOTEM) in Pediatric Patients With Relapsed or Refractory Neuroblastoma and Other Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study halted early due to high toxicity risk (from BHLRM model) in combo treatment and inability to identify recommended Phase 2 dose in initial phase (Phase 1-Part A), making continuation to subsequent phases (Phase 1-Part B and Phase 2) unfeasible.
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Innovative Therapies For Children with Cancer Consortium (Other)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CLEE011Q12101; 2024-512095-35-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2022-06-17; First posted 2022-06-23 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Neuroblastoma
Keywords: neuroblastoma; medulloblastoma; high-grade glioma; malignant rhabdoid tumors; rhabdomyosarcoma; relapsed; refractory; pediatric
MeSH Terms: conditions — Neuroblastoma; Medulloblastoma; Glioma; Rhabdomyosarcoma; Recurrence | interventions — Topotecan; Temozolomide; ribociclib

STUDY DESIGN:
Intervention Model Description: Cohort A1 - concurrent regimen Cohort A2 - sequential regimen Cohort A3 (post protocol amendment #2) - concurrent
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Phase I-part A: Ribociclib + Topotecan and Temozolomide (Experimental): Participants with r/r NB, MB, HGG, MRT or RMS will be treated with ribociclib in combination with topotecan and temozolomide to determine MTD and/or RP2D. Ribociclib dose will be escalated with topotecan and temozolomide.
  Interventions: Drug: Topotecan; Drug: Temozolomide; Drug: Ribociclib

INTERVENTIONS:
Drug: Topotecan — Starting out dose of topotecan administered at standard dose given to neuroblastoma patients (0.75 mg/m2/day).
  Other Names: Hycamtin
Drug: Temozolomide — Starting out dose of temozolomide for cohort A1 and A2 for Phase 1-Part A: 150mg/m2/day. Starting out dose for subsequent cohorts, Cohort A3 and onwards, in Phase 1-Part A will initiate at 100mg/m2/day.
  Other Names: Temodar
Drug: Ribociclib — Starting out dose of ribociclib for cohort A1 Phase 1-Part A: 200mg/m2/day. Starting out dose for Cohort A2 and A3 was 100mg/m2/day.
  Other Names: Kisqali; LEE011

SUMMARY:
This is a Phase I/II study to assess the efficacy and safety of ribociclib in combination with topotecan and temozolomide (TOTEM) in pediatric patients with relapsed or refractory (r/r) neuroblastoma (NB), and other solid tumors, including medulloblastoma (MB), high-grade glioma (HGG), malignant rhabdoid tumors (MRT), and rhabdomyosarcoma (RMS).

DETAILED DESCRIPTION:
The study is structured into two parts: Phase I - Part A (dose finding) and Phase I - Part B (multiple expansion cohorts). Phase II may commence following the evaluation of Phase I data, which includes safety, tolerability, efficacy, pharmacokinetics, and biomarker data. Additionally, other emerging data that could influence the treatment landscape will be considered before initiating Phase II in patients with relapsed or refractory neuroblastoma (NB) and/or other tumors studied in Phase I.

- Phase I - Part A (dose finding): This phase aims to determine the maximum tolerated dose (MTD) and/or the recommended Phase II dose (RP2D) of ribociclib in combination with TOTEM.

Due to the early termination of the trial, Phase I - Part B (multiple expansion cohorts) and Phase II (double-blind, randomized, placebo-controlled in relapsed or refractory NB) were not initiated.

ELIGIBILITY:
Inclusion Criteria:

1. Participants and/or guardian have the ability to understand and the willingness to sign a written informed consent document.
2. Age ≥ 12 months and ≤ 21 years at the time of signing consent form Note: The first dose level of Phase I - part A (dose finding) will enroll participants ≥ 12 years - 21 years old, and may expand to younger participants (≥ 12 months to < 12 years) as determined by the data.
3. Histologically or cytologically confirmed solid tumors listed below that have progressed despite standard therapy or for which no effective standard therapy exists.

   1. Neuroblastoma (for Phase I and Phase II): Histologically proven neuroblastoma as per International Neuroblastoma Staging System (INSS); Relapsed or refractory disease; Measurable disease per International Neuroblastoma Response criteria (INRC); Bone marrow only disease not eligible; Available MYCN status before screening
   2. Medulloblastoma (for Phase I) regardless of genetic status (i.e. Groups 3 or 4 WNT-activated or non-WNT, SHH-activated or non-SHH)
   3. High-grade glioma (for Phase I): including HGG NOS, WHO Grade III or Grade IV; Glioblastoma, IDH-wildtype or IDH-mutant; Anaplastic astrocytoma, IDH-mutant; Anaplastic oligodendroglioma, IDH-mutant; Anaplastic pleomorphic xanthoastrocytoma; Diffuse midline gliomas, H3 K27-altered; Diffuse hemispheric glioma, H3 G34-mutant; Diffuse pediatric-type HGG, H3-wildtype and IDH-wildtype.
   4. Malignant rhabdoid tumor (for Phase I) includes diagnoses of atypical teratoid/rhabdoid tumor (AT/RT), and rhabdoid tumor of the kidney (RTK), and other soft tissues as defined by 2 of the 3 following criteria; either (1)+(2) or (1)+(3): (1) Morphology and immunophenotypic panel consistent with rhabdoid tumor; (2) Loss of SMARCB1 confirmed by immunohistochemistry; (3) Molecular confirmation of tumor-specific bi-allelic SMARCB1 loss/mutation is encouraged in cases where SMARCB1 immunohistochemistry is equivocal, and required if SMARCB1 immunohistochemistry is not available
   5. Rhabdomyosarcoma (for Phase I) independent of fusion status and subtype
4. Participants with CNS disease who are on corticosteroids should take stable doses for at least 7 days prior to first dose of ribociclib with no plans for escalation.
5. Performance status:

   1. ≤ 16 years: Lansky Play score ≥ 50%
   2. >16 years: Karnofsky performance status ≥ 50% or ECOG < 3
6. Life expectancy of ≥ 12 weeks at the time of enrollment
7. Adequate bone marrow function (bone marrow may be involved with tumor) and organ function
8. Adequate hepatic, renal, cardiac function
9. Females who are sexually active must agree to use highly effective contraception during and for 6 months after treatment. Additionally, females of childbearing potential must have a negative serum pregnancy test within 7 days prior to the first dose of study medication. Pregnant or lactating females are not eligible for the study.
10. Sexually active males (including those that have had a vasectomy), who do not agree to abstinence, must be willing to use a condom during intercourse while on study treatment and for 6 months after stopping treatment.

Exclusion Criteria:

1. Known hypersensitivity to any of the excipients of ribociclib or topotecan or temozolomide.
2. Not recovered from clinical and laboratory acute toxicities related to prior anti-cancer therapies
3. Concurrent severe and/or uncontrolled concurrent medical conditions (serious infections or significant cardiac, pulmonary, hepatic, psychiatric, GI disease, or other organ dysfunction) that in the investigator's judgement could compromise their ability to tolerate or absorb protocol therapy or would interfere with the study procedures or results
4. Clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormality
5. History of QTc prolongation; taking medications with a known risk to prolong the QT interval hat cannot be discontinued or replaced by safe alternative medication
6. Currently taking medications that are mainly metabolized by CYP3A4/5 with a narrow therapeutic index, strong inducers or inhibitors of CYP3A4/5, herbal preparations/medications and dietary supplements
7. Vaccinated with live, attenuated vaccines within 4 weeks
8. Participated in a prior investigational study within 30 days
9. Received prior treatment with a CDK4/6 inhibitor
10. Received last dose of anticancer therapy (including experimental) within 4 weeks
11. Previous myeloablative therapy with autologous hematopoietic stem cell rescue within 8 weeks
12. Allogeneic stem cell transplant within 3 months
13. Has last fraction of radiation within 4 weeks
14. Major surgery within 2 weeks
15. Pregnant or nursing (breast feeding) female participant or female participant who plans to become pregnant or breast-feed during the trial.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 12 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2022-12-27 (Actual); Primary Completion 2025-02-26 (Actual); Study Completion 2025-02-26 (Actual)

PRIMARY OUTCOMES:
Phase 1- Part A: Percentage of participants with Dose Limiting Toxicities (DLTs) in Cycle 1 | Up to 28 days
  Percentage of participants with DLTs during first cycle of treatment (each cycle is 28 days) for each dose level associated with administration of ribociclib in combination with topotecan and temozolomide.
  A DLT is defined as an adverse event or abnormal laboratory value suspected to be related with study treatment.

SECONDARY OUTCOMES:
Plasma concentrations of ribociclib (Phase I-Part A) | Cycle 1 day 1 and 15; Cycle 2 Day 15. Cycle=28 days
  Pharmacokinetic (PK) blood samples will be collected at selected time-points to determine ribociclib plasma concentrations from participants in Phase I-Part A, Phase I-Part B and Phase II
Area under the plasma concentration-time curve (AUC) of ribociclib (Phase I-Part A) | Cycle 1 day 1 and 15; Cycle 2 Day 15. Cycle=28 days
  PK blood samples will be collected at selected time-points to determine AUC of ribociclib from participants in Phase I-Part A, Phase I-Part B and Phase II
Maximum plasma concentration (Cmax) of ribociclib (Phase I-Part A) | Cycle 1 day 1 and 15; Cycle 2 Day 15. Cycle=28 days
  PK blood samples will be collected at selected time-points to determine Cmax of ribociclib from participants in Phase I-Part A, Phase I-Part B and Phase II
Time of maximum plasma concentration (Tmax) of ribociclib (Phase I-Part A) | Cycle 1 day 1 and 15; Cycle 2 Day 15. Cycle=28 days
  PK blood samples will be collected at selected time-points to determine Cmax of ribociclib from participants in Phase I-Part A and Phase I-Part B.
Percentage of participants with dose interruptions and dose reductions (Phase I-Part A) | Up to 12 months
  Percentage of participants with dose interruptions and dose reductions for participants in Phase I-Part A, Phase I-Part B and Phase II

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (6):
- United States (3):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Cohen Children's Medical Center of New York, New Hyde Park, New York
  - St Jude s Childrens Research Hospital, Memphis, Tennessee
- Novartis Investigative Site, Cologne, Germany
- Novartis Investigative Site, Milan, MI, Italy
- Novartis Investigative Site, Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.

REFERENCES:
- See also: Link to study results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18345
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2787